CLINICAL TRIAL: NCT01096394
Title: Orthotopic Propagation of Primary Human Ovarian Tumors for Preclinical Investigation of Novel Anti-Tumor Agents.
Brief Title: Collection of Tissue Samples From Patients With Stage III or Stage IV Ovarian Epithelial Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Dineo Khabele, Assistant Professor, Vanderbilt University
Other Study IDs: 090075; P30CA068485 (NIH); VU-VICC-GYN-0917 (Other: Vanderbilt Ingram Cancer Center); IRB# 090075 (Other: Vanderbilt University Human Protections Program)
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Metastatic and primary tumor tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ovarian cancer: Patients with presumed Stage III-IV ovarian, primary fallopian tube, or primary peritoneal papillary serous carcinoma.

SUMMARY:
RATIONALE: Collecting and storing samples of tumor tissue and ascites fluid from patients to test in the laboratory may help the study of cancer.

PURPOSE: This pre-clinical research study is collecting tissue samples and ascites fluid from patients with stage III or stage IV ovarian/primary peritoneal/fallopian tube epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To generate a translational ovarian cancer model using tumor tissue and cells from patients with stage III-IV ovarian/primary peritoneal/fallopian tube epithelial cancer for drug response and development.

OUTLINE: Tissue and fluid samples are collected at the time of surgery or paracentesis and used in laboratory experiments and in animal models. Health data is collected from patient medical records before, during, and after surgery.

After surgery, patients are followed up for 5 years.

ELIGIBILITY:
INCLUSION:

• Females age 18-80 with a diagnosis of Stage III-IV ovarian cancer, primary fallopian tube, or primary peritoneal papillary serous carcinoma and scheduled treatment for epithelial ovarian malignancies.

EXCLUSION:

* Patients with less than Stage III epithelial ovarian cancer, primary fallopian tube, or primary peritoneal papillary serous carcinoma
* Patients who have received prior chemotherapy
* Patients who have nonepithelial ovarian cancer, primary fallopian tube, or primary peritoneal carcinoma
* Patients who have malignancy other than ovarian cancer, primary fallopian tube, or primary peritoneal carcinoma

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females age 18-80 with a diagnosis of Stage III-IV ovarian cancer, primary fallopian tube, or primary peritoneal papillary serous carcinoma and scheduled treatment for epithelial ovarian malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Establishment of a "live" library of primary ovarian epithelial tumors | 5 year follow up of outcome.
  Our approach is to establish a "live" library of primary tumors from patients diagnosed with ovarian cancer by transplanting this tissue into a host mouse model. This preclinical model system will allow us to test the response to standard and novel therapeutics and will provide a perpetual tumor archive for future experiments that will probe critical molecular pathways involved in the pathogenesis of ovarian cancer and similar cancer types (primary peritoneal and fallopian tube).

CONTACTS AND LOCATIONS:
Overall Officials: Dineo Khabele, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States